CLINICAL TRIAL: NCT04940793
Title: Visual and Refractive Outcomes of a New Diffractive Trifocal Toric Intraocular Lens
Acronym: RibeiroPODFT
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ribeiro - POD FT
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Cataract
Keywords: Trifocal; Toric; Hydrophilic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients indicated for cataract surgery who are candidates for a trifocal IOL implantation and have corneal astigmatism over 1.00 D will be selected for inclusion by the investigators
  Interventions: Device: POD FT

INTERVENTIONS:
Device: POD FT — Cataract surgery

SUMMARY:
The purpose of this study is to investigate the visual performance and refractive predictability with the diffractive toric Finevision POD FT IOL. Predicted and achieved visual outcomes, visual performance at near, intermediate and far distance as well as photic phenomena, rotational stability and spectacle independence will be investigated. The follow-up period is 3 months after which vision and refraction should have stabilized.

DETAILED DESCRIPTION:
This prospective study was performed to investigate the visual performance and refractive predictability with the diffractive toric Finevision POD FT IOL (PhyslOL, Belgium). Predicted and achieved visual outcomes, visual performance at near, intermediate and far distance as well as rotational stability have been analyzed. The follow-up period was 6 months. All IOL implantations were performed by the investigators Dr. Filomena Ribeiro and Dr. Tiago B Ferreira (Hospital da Luz, Lisboa, Portugal). The study population consists of patients undergoing routine cataract surgery. The study patients underwent binocular implantation of Finevision IOLs depending on the preoperative amount of corneal astigmatism (either a toric POD FT IOL in both eyes or a POD FT in the study eye and a non-toric POD F IOL in the contralateral eye).

ELIGIBILITY:
Inclusion Criteria:

* age 21 and older
* bilateral implantation of a Finevision trifocal diffractive IOL (either a POD FT in both eyes or a POD FT in the study eye and a POD F in the contralateral eye)
* bilateral cataract surgery with grade 1-4 cataract
* regular corneal astigmatism of 1.00 D or more before surgery in the study eye
* previous written informed consent to surgery. Written informed consent to participation in the study and data protection

Exclusion Criteria:

* relevant concomitant ophthalmic diseases (such as pseudoexfoliation, glaucoma, traumatic cataract and other co-morbidity that could affect capsular bag stability (e.g. Marfan syndrome)
* irregular corneal astigmatism, any abnormality in corneal topography
* systemic disease with impact on visual outcome
* disability to understand and/or fill in patient questionnaires
* history of other relevant previous ocular surgery (such as corneal surgery, glaucoma surgery, vitreoretinal surgery) which might affect capsular stability or visual outcomes
* expected residual cylinder ≥ 0.50 D

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients indicated for cataract surgery who are candidates for a trifocal IOL implantation and have corneal astigmatism over 1.00 D will be selected for inclusion by the investigators. Only patients with binocular implantation of a Finevision IOL will be included (either a POD FT in both eyes or a POD FT in the study eye and a POD F in the contralateral eye).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Visual performance | 3 Months
  The purpose of this study is to investigate the visual performance of the diffractive toric Finevision POD FT IOL.
Refractive predictability | 3 Months
  The purpose of this study is to investigate the refractive predictability of the diffractive toric Finevision POD FT IOL.

SECONDARY OUTCOMES:
Visual performance : predicted and achieved | 3 Months
  The purpose of this study is to investigate the visual performance of the diffractive toric Finevision POD FT IOL. Predicted and achieved visual outcomes will be investigated.
Visual performance at near, intermediate and far distance | 3 Months
  The purpose of this study is to investigate the visual performance of the diffractive toric Finevision POD FT IOL. Visual performance at near, intermediate and far distance will be investigated.
Refractive predictability: photic phenomena | 3 Months
  The purpose of this study is to investigate the refractive predictability of the diffractive toric Finevision POD FT IOL. The photic phenomena will be investigated.
Refractive predictability: rotational stability | 3 Months
  The purpose of this study is to investigate the refractive predictability of the diffractive toric Finevision POD FT IOL. The rotational stability will be investigated.
Refractive predictability: spectacle independence | 3 Months
  The purpose of this study is to investigate the refractive predictability of the diffractive toric Finevision POD FT IOL. The spectacle independence will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Filomena Ribeiro, MD, PhD, FEBO, Principal Investigator — Hospital da Luz
Locations (1):
- Hospital da Luz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Visser N, Bauer NJ, Nuijts RM. Toric intraocular lenses: historical overview, patient selection, IOL calculation, surgical techniques, clinical outcomes, and complications. J Cataract Refract Surg. 2013 Apr;39(4):624-37. doi: 10.1016/j.jcrs.2013.02.020. PMID 23522584
- [Result] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Result] Wolffsohn JS, Jinabhai AN, Kingsnorth A, Sheppard AL, Naroo SA, Shah S, Buckhurst P, Hall LA, Young G. Exploring the optimum step size for defocus curves. J Cataract Refract Surg. 2013 Jun;39(6):873-80. doi: 10.1016/j.jcrs.2013.01.031. PMID 23688874
- [Result] Vryghem JC, Heireman S. Visual performance after the implantation of a new trifocal intraocular lens. Clin Ophthalmol. 2013;7:1957-65. doi: 10.2147/OPTH.S44415. Epub 2013 Oct 1. PMID 24124348
- [Result] Sheppard AL, Shah S, Bhatt U, Bhogal G, Wolffsohn JS. Visual outcomes and subjective experience after bilateral implantation of a new diffractive trifocal intraocular lens. J Cataract Refract Surg. 2013 Mar;39(3):343-9. doi: 10.1016/j.jcrs.2012.09.017. Epub 2013 Jan 16. PMID 23332118
- [Result] Cochener B, Vryghem J, Rozot P, Lesieur G, Heireman S, Blanckaert JA, Van Acker E, Ghekiere S. Visual and refractive outcomes after implantation of a fully diffractive trifocal lens. Clin Ophthalmol. 2012;6:1421-7. doi: 10.2147/OPTH.S32343. Epub 2012 Sep 3. PMID 22969289
- [Result] Roensch MA, Charton JW, Blomquist PH, Aggarwal NK, McCulley JP. Resident experience with toric and multifocal intraocular lenses in a public county hospital system. J Cataract Refract Surg. 2012 May;38(5):793-8. doi: 10.1016/j.jcrs.2011.11.043. Epub 2012 Mar 15. PMID 22425363
- [Result] Visser N, Nuijts RM, de Vries NE, Bauer NJ. Visual outcomes and patient satisfaction after cataract surgery with toric multifocal intraocular lens implantation. J Cataract Refract Surg. 2011 Nov;37(11):2034-42. doi: 10.1016/j.jcrs.2011.05.041. Epub 2011 Sep 22. PMID 21940140
- [Result] Bellucci R, Bauer NJ, Daya SM, Visser N, Santin G, Cargnoni M, Nuijts RM; Lisa Toric Study Group. Visual acuity and refraction with a diffractive multifocal toric intraocular lens. J Cataract Refract Surg. 2013 Oct;39(10):1507-18. doi: 10.1016/j.jcrs.2013.04.036. PMID 24075158
- [Result] Alfonso JF, Knorz M, Fernandez-Vega L, Rincon JL, Suarez E, Titke C, Kohnen T. Clinical outcomes after bilateral implantation of an apodized +3.0 D toric diffractive multifocal intraocular lens. J Cataract Refract Surg. 2014 Jan;40(1):51-9. doi: 10.1016/j.jcrs.2013.06.026. PMID 24355720
- [Result] Ferreira TB, Marques EF, Rodrigues A, Montes-Mico R. Visual and optical outcomes of a diffractive multifocal toric intraocular lens. J Cataract Refract Surg. 2013 Jul;39(7):1029-35. doi: 10.1016/j.jcrs.2013.02.037. Epub 2013 May 13. PMID 23680631
- [Result] Knorz MC, Rincon JL, Suarez E, Alfonso JF, Fernandez-Vega L, Titke C, Kohnen T, Tucker S. Subjective outcomes after bilateral implantation of an apodized diffractive +3.0 D multifocal toric IOL in a prospective clinical study. J Refract Surg. 2013 Nov;29(11):762-7. doi: 10.3928/1081597X-20131021-06. PMID 24203808
- [Result] Chassain C, Pagnoulle C, Gobin L, Rozema J. [Evaluation of a new intraocular lens platform: centration and rotational stability]. J Fr Ophtalmol. 2013 Apr;36(4):336-42. doi: 10.1016/j.jfo.2012.04.012. Epub 2013 Jan 24. French. PMID 23352708